CLINICAL TRIAL: NCT00542607
Title: Trial to Compare the Efficacy and Safety of Levocetirizine 5 mg od and Fexofenadine 120 mg od in Reducing Symptoms of Seasonal Allergic Rhinitis in Grass Pollen Sensitized Adults
Brief Title: Efficacy and Safety of Levocetirizine and Fexofenadine in Reducing Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A00324
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levocetirizine dihydrochloride

SUMMARY:
No information was yet available over the effect of levocetirizine in children under 12 years. The aim of this double-blind, placebo-controlled study was to assess the efficacy and safety of levocetirizine in children from 6 to 12 years old with perennial allergic rhinitis due to house dust mites.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 to 55 years both inclusive
* suffering at least 2 years of seasonal allergic rhinitis due to grass pollen
* positive RAST and/or positive skin prick test
* comply with study restrictions

Exclusion Criteria:

* known alcohol or drug addiction or abuse
* known allergy/intolerance to lactose, cellulose, cornstarch
* presence of nasal anatomical deformities leading to > 50% obstruction
* ENT infection within 30 days of the study
* use of disallowed medication
* ongoing desensitization
* known cardiac, renal or hepatic dysfunction
* presenting allergic bronchial asthma
* use of cimetidine
* intending to donate blood during the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2002-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the mean Major symptom complex score over the last 2 hours of a 24-hour coverage

SECONDARY OUTCOMES:
The change from baseline of the mean MSC score over time interval 3
the change from baseline of the mean MSC score over time intervals 1 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: UCb Clinical Trial Call Center, Study Director — UCB Pharma